CLINICAL TRIAL: NCT00068146
Title: Study of Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) for the Evaluation of the Autoimmune Lymphoproliferative Syndrome (ALPS) and ALPS-Associated Lymphoma
Brief Title: Fluorodeoxyglucose-Positron Emission Tomography (FDG-PET) to Evaluate Autoimmune Lymphoproliferative Syndrome (ALPS) and ALPS-associated Lymphoma
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020308; 02-I-0308
Record Dates: First submitted 2003-09-09; First posted 2003-09-09 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-11-26

CONDITIONS: Lymphoproliferative Disorders; Lymphoma
Keywords: Adenopathy; Genetic Disorder; Apoptosis; Diagnostic Imaging; Hodgkins; Autoimmune Lymphoproliferative; Syndrome; ALPS; ALPS-Associated Lymphoma
MeSH Terms: conditions — Lymphoproliferative Disorders; Lymphoma; Lymphadenopathy; Genetic Diseases, Inborn; Syndrome

SUMMARY:
This study will evaluate the usefulness of FDG-PET scanning in distinguishing autoimmune lymphoproliferative syndrome (ALPS) from lymphoma. Lymphoma is cancer of the lymph system. ALPS is a condition involving persistent enlargement of the lymph glands, spleen, or liver, and a range of other problems relating to blood cell counts and abnormal immune activity, in which the immune system attacks healthy tissues. People with ALPS particularly those with an abnormal Fas gene also have an increased risk of developing lymphoma. The Fas gene codes for a protein that causes immune cells called lymphocytes to die when they are no longer needed.

FDG-PET is a new nuclear imaging test that is very effective in detecting lymphoma. It is important to identify these cancers as quickly as possible, since some are very curable when caught early. Since ALPS and lymphoma share several common characteristics, a reliable, non-invasive method of distinguishing the two, such as FDG-PET might offer, is crucial. FDG-PET uses a radioactive sugar molecule to produce images that show the metabolic activity of tissues. Because cancer cells grow and divide more rapidly than normal cells, they metabolize more sugar for fuel. This increased activity identifies them as cancer in FDG-PET scanning. For this procedure, the subject is injected with the sugar molecule and lies in a doughnut-shaped machine (PET camera) for the imaging.

Adults and children 10 years old or older with ALPS, with or without lymphoma, may be eligible for this study. Candidates will be screened with a physical examination, blood tests, and computed tomography (CT) scan.

Participants will have an FDG-PET scan and a DEXA scan. The DEXA scan measures fat and non-fat tissue and is used help interpret the FDG-PET results. For this test, the subject lies on a table while a fast X-ray is taken from head to toe.

Patients who develop signs or symptoms suggesting the development or recurrence of lymphoma (such as further enlargement of lymph glands, unexplained fever or weight loss, or abnormal scans) may undergo a tissue biopsy. For this procedure, a small piece of lymph or other tissue is surgically removed for examination under the microscope. In addition, patients who develop these symptoms may be asked to undergo additional FDG-PET scans up to two a year in patients without lymphoma, and as many as needed in patients with lymphoma to evaluate their response to treatment and guide future therapy.

DETAILED DESCRIPTION:
The Autoimmune Lymphoproliferative Syndrome (ALPS) is an inherited disorder associated with defective lymphocyte apoptosis, which is clinically characterized by prominent non-malignant lymphadenopathy, hepatosplenomegaly and overt autoimmune diseases such as hemolytic anemia, autoimmune thrombocytopenia and neutropenia. Additionally, ALPS patients have a significantly increased risk of developing non-Hodgkin's and Hodgkin's lymphoma.

The diagnosis of lymphoma is particularly troublesome in ALPS because many ALPS manifestations overlap with clinical features suggestive of lymphoma. Therefore, individuals with ALPS may undergo repeated biopsies during the course of the disease. Finding a non-invasive test that can predictably discriminate benign from malignant lymphadenopathy in ALPS, and that can help discern whether a more invasive lymph node biopsy is necessary, would be very desirable.

Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) is an increasingly used non-invasive imaging technique for staging and monitoring therapeutic responses in patients with lymphoma. This technique might be able to assist us in distinguishing whether enlargement of lymph nodes is due to ALPS versus ALPS associated lymphoma. However, FDG-PET has not been studied in patients with ALPS. This study will first explore whether ALPS patients with lymphadenopathy show FDG uptake. If uptake is shown, the study will obtain initial quantitative data to compare FDG uptake in ALPS patients with lymphadenopathy, and ALPS patients with associated lymphoma. The ultimate goal is to assess FDG-PET as a reliable non-invasive method to differentiate lymphadenopathy due to ALPS versus that of ALPS associated lymphoma.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALPS Patients without Lymphoma:

Participants must:

1. Fulfill current criteria for the diagnosis of ALPS as follows:

   1. Documented chronic nonmalignant lymphadenopathy and/or splenomegaly, and
   2. Greater than or equal to 1.5 percent TCR alpha/beta+ CD4- CD8- T cells in the peripheral blood.
2. Be enrolled in ALPS Natural History Protocol 93-I-0063.
3. Have clinical evidence of lymphadenopathy as defined by multiple palpable lymph nodes of at least 1cm or radiographic evidence of lymphadenopathy as defined by multiple lymph nodes of at least 1 cm on CT scan, during an evaluation at the NIH Clinical Center.
4. Be 8 years of age or older. The study will be targeted to children 8 years of age or older and adults because younger children may not be able to stay still for the duration of the FDG-PET scan procedure. Sedation will not be used in children in this study, except for clinically indicated procedures such as FDG-PET scans in children with lymphoma.
5. Be due for their routine [every 2 years] CT scan under protocol 93-I-0063, or be in need of a CT scan for medical reasons [e.g. marked change in adenopathy]. CT scan within 3 months prior to FDG-PET scan is necessary to locate the nodes for appropriate FDG-PET analysis.

ALPS Patients with Lymphoma:

Patients must:

1. Fulfill current criteria for the diagnosis of ALPS as follows:

   1. Documented chronic nonmalignant lymphadenopathy and/or splenomegaly.
   2. Greater than or equal to 1.5 percent TCR alpha/beta + CD4- CD8 -T cells in the peripheral blood.
2. Be enrolled in ALPS Natural History Protocol 93-I-0063.
3. Have a histologically proven diagnosis of lymphoma, confirmed by the Laboratory of Pathology, NCI (Anatomic Pathology Dept, CC) whether yet treated or not. Lymphomas will be classified according to the WHO classification, using appropriate immunophenotypic and histological features.

EXCLUSION CRITERIA:

1. Patient will be excluded if any of the following are present:
2. Concurrent infection or inflammatory disease (e.g., sarcoidosis), which itself often shows increased FDG uptake by PET and which could interfere with the interpretation of study results.
3. Active neoplasia other than lymphoma.
4. History of chemotherapy or radiation treated malignancy within 5 years prior to study procedure, except for lymphoma.
5. Hyperglycermia (regardless of etiology) determined by fasting glucose of greater than 130 mg/dl. Individual with an underlying defect of glucose metabolism may exhibit abnormal metabolism of FDG.
6. Weights in excess of 136 kg, which will exceed the weight limit for the scanner table.
7. Pregnancy and breast-feeding. For women of childbearing potential, a negative urine or serum pregnancy test is required within 24 hours prior to an FDG-PET scan.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2002-09-19; Study Completion 2012-11-26

CONTACTS AND LOCATIONS:
Overall Officials: V. Koneti Rao, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sneller MC, Wang J, Dale JK, Strober W, Middelton LA, Choi Y, Fleisher TA, Lim MS, Jaffe ES, Puck JM, Lenardo MJ, Straus SE. Clincal, immunologic, and genetic features of an autoimmune lymphoproliferative syndrome associated with abnormal lymphocyte apoptosis. Blood. 1997 Feb 15;89(4):1341-8. PMID 9028957
- [Background] Straus SE, Sneller M, Lenardo MJ, Puck JM, Strober W. An inherited disorder of lymphocyte apoptosis: the autoimmune lymphoproliferative syndrome. Ann Intern Med. 1999 Apr 6;130(7):591-601. doi: 10.7326/0003-4819-130-7-199904060-00020. PMID 10189330
- [Background] Avila NA, Dwyer AJ, Dale JK, Lopatin UA, Sneller MC, Jaffe ES, Puck JM, Straus SE. Autoimmune lymphoproliferative syndrome: a syndrome associated with inherited genetic defects that impair lymphocytic apoptosis--CT and US features. Radiology. 1999 Jul;212(1):257-63. doi: 10.1148/radiology.212.1.r99jl40257. PMID 10405750